CLINICAL TRIAL: NCT02452840
Title: Adjunctive Photodynamic Therapy for Persistent Disease Activity in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Photodynamic Therapy for PDA in NV AMD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00057705
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Neovascular Age-related Macular Degeneration; Macular Degeneration
Keywords: neovascular age-related macular degeneration; anti-vascular endothelial growth factor; verteporfin; photodynamic therapy; persistent disease activity
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NVAMD Patients with PDA: NVAMD Patients with PDA
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this prospective observational study is to assess the potential clinical effects of adjunctive verteporfin photodynamic therapy (PDT) for persistent disease activity among patients with neovascular age-related macular degeneration (NV AMD). No specific interventions will occur as part of the study; participating subjects undergoing PDT as part of standard-of-care will be asked to consent to prospective collection of data from their medical records for up to five years from the date of consent, including results from ophthalmologic exams, imaging, and treatments. The primary study outcome will be the percentage of subjects with resolution of persistent disease activity at six months post-PDT treatment. Aside from a small risk of loss of confidentiality, risks associated with this study are no greater than those related to standard of care.

DETAILED DESCRIPTION:
NV AMD remains the leading cause of vision loss among people over 65. Intravitreal injections with drugs that block vascular endothelial growth factor (VEGF), a major protein mediator of angiogenesis and vascular leakage, have revolutionized treatment of NV AMD. However, less than 40% of treated patients have clinically significant improvement in vision. Further, in spite of continuous monthly anti-VEGF therapy, up to 40-50% of patients demonstrate persistent disease activity (PDA), defined as (1) unresolved intraretinal, subretinal, or sub-retinal pigment epithelium fluid; (2) progressive lesion enlargement and fibrosis; and/or (3) persistent or new hemorrhage, assessed after either loading dose therapy or after sustained treatment with anti-VEGF. Since affected patients are at increased risk for long-term vision loss, PDA remains a vital clinical unmet need.

Verteporfin PDT (Visudyne®, Bausch+Lomb) was approved over 10 years ago by the FDA for treatment of NV AMD, prior to the advent of anti-VEGF therapy. As a monotherapy, PDT is much less effective than anti-VEGF therapy in improving vision for NV AMD patients. Furthermore, in general, PDT in combination with anti-VEGF therapy does not offer benefit over anti-VEGF therapy alone, when assessed among previously treatment-naïve NV AMD patients. However, it is unknown whether adjunctive PDT may be effective for the treatment of PDA. The investigators have performed several retrospective studies of PDA and adjunctive PDT among NV AMD patients in the Duke Medical Retina practice. Preliminary results indicate that moderate to severe PDA occurs in over 40% of NV AMD patients, and that adjunctive verteporfin PDT may be effective in improving PDA and vision for affected patients.

The present study will assess potential clinical benefits of adjunctive PDT for NV AMD patients with PDA in spite of anti-VEGF therapy in a prospective observational clinical case series.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NV AMD
* Evidence of PDA in spite of loading dose intravitreal anti-VEGF therapy. PDA is defined as (1) unresolved intraretinal, subretinal, or sub-retinal pigment epithelium fluid; (2) progressive lesion enlargement and fibrosis; and/or (3) persistent or new hemorrhage.
* Undergoing adjunctive verteporfin PDT for the treatment of PDA
* Able to give written informed consent

Exclusion Criteria:

* Prior PDT treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NVAMD with evidence of PDA in spite of loading dose intravitreal anti-VEGF therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with resolution of PDA | Six months post-PDT treatment

SECONDARY OUTCOMES:
Mean change in best-corrected ETDRS visual acuity from baseline | Six months post-PDT treatment
Percentage of subjects with 2-line ETDRS visual acuity gain from baseline | Six months post-PDT treatment
Percentage of subjects with 2-line ETDRS visual acuity loss from baseline | Six months post-PDT treatment
Mean change in central foveal thickness by SD-OCT from baseline | Six months post-PDT treatment
Mean change in choroidal neovascularization lesion size by fluorescein angiography from baseline | Six months post-PDT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cousins, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States